CLINICAL TRIAL: NCT06921265
Title: Tailored Neuromodulation Intervention to Enhance Speech and Language Training in Patients With Primary Progressive Aphasia: EEG and MRI Targeted Transcranial Magnetic Stimulation
Brief Title: Targeted Transcranial Magnetic Stimulation to Improve Language and Speech in Patients With Primary Progressive Aphasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Prof., Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEUROTECH_002_PPA
Record Dates: First submitted 2025-03-05; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Primary Progressive Aphasia(PPA)
Keywords: Non-Invasive Brain Stimulation; blood sample; Non - Fluent Variant Primary Progressive Aphasia (nfvPPA); Primary Progressive Aphasia (PPA); Speak and Language Therapy (SLT); Functional Magnetic Resonance Imaging (fMRI); electroencephalogram (EEG); Functional Near Infrared Spectroscopy (fNIRS); Semantic Variant Primary Progressive Aphasia (svPPA); Logopenic Variant Primary Progressive Aphasia (lvPPA)
MeSH Terms: conditions — Aphasia, Primary Progressive; Speech | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Training with SLT (Active Comparator): The training will be tailored to each PPA variant. svPPA and lvPPA will undergo the LRC training, while nfvPPA will undergo the VISTA training.
  Interventions: Behavioral: Training with Speech Language Therapy
- SLT + Brain STIM (Standard rTMS + targeted rTMS) (Experimental): Patients will perform the same exercises as SLT group, combined with brain STIM. The SLT + non invasive brain STIM (standard rTMS + targeted rTMS) group will undergo 2 cycles of 6-week training, separated by a 12-week washout period with a cross-over design, according to a randomization procedure.
  Half of subjects will first receive 6-week SLT training + standard rTMS followed by 6-week SLT training associated with targeted rTMS, according to the crossover design.
  Interventions: Behavioral: Training with Speech Language Therapy; Device: Standard rTMS; Device: Targeted rTMS; Device: Standard rTMS (first cycle); Device: Targeted rTMS (second cycle)
- Healthy controls (No Intervention): Age- and sex-matched healthy subjects recruited to compare neuropsychological, functional magnetic resonance imaging and neurophysiological characteristics at baseline
- Experimental: SLT + Brain STIM (targeted rTMS + Standard rTMS) (Experimental): Patients will perform the same exercises as SLT group, combined with non invasive brain STIM. The SLT + STIM (targeted rTMS + standard rTMS) group will undergo 2 cycles of 6-week training, separated by a 12-week washout period with a cross-over design, according to a randomization procedure. Half of subjects will first receive 6-week SLT training + targeted rTMS followed by 6-week SLT training associated with standard rTMS, according to the crossover design.
  Interventions: Behavioral: Training with Speech Language Therapy; Device: Standard rTMS; Device: Targeted rTMS; Device: Standard rTMS (second cycle); Device: Targeted rTMS (first cycle)

INTERVENTIONS:
Behavioral: Training with Speech Language Therapy — The SLT will consist of an online intervention performed through a web-based platform.
  The SLT training of the SLT group will consist of 2 cycles of training lasting 1 (rest) + 5 (training) weeks, 3 times per week, 1 hour each session, separated by a 12-week washout period.
  Arms: Experimental: SLT + Brain STIM (targeted rTMS + Standard rTMS); SLT + Brain STIM (Standard rTMS + targeted rTMS); Training with SLT
Device: Standard rTMS — Stimulation of DLPFC; rTMS will be administered as high-frequency (20Hz) in 2 second trains (40 pulses per train) with an inter-train interval of 22 seconds for a total of 50 trains (2000 pulses per session) at 120% of the patient's resting motor threshold. Patients will undergo an induction with 20-minutes rTMS protocol for 5 consecutive days, then they will start a maintenance phase where rTMS will be performed 3 days a week per 20 minutes preceding the SLT session, for a total of 20 sessions (of whom 15 combined with SLT).
  Arms: Experimental: SLT + Brain STIM (targeted rTMS + Standard rTMS); SLT + Brain STIM (Standard rTMS + targeted rTMS)
Device: Targeted rTMS — The protocol will be the same as standard STIM. The site of stimulation will be defined using EEG/fMRI recordings of language tasks (syntax production for nfvPPA; silent naming for svPPA and lvPPA) to evidence the areas of higher activation/connectivity of the language network. We will define the area of higher fMRI activation; then, we will use fMRI-EEG connectivity and spectral activity to select the site of stimulation, among the areas with the highest fMRI activation and the highest Beta/Gamma frequencies.
  Arms: Experimental: SLT + Brain STIM (targeted rTMS + Standard rTMS); SLT + Brain STIM (Standard rTMS + targeted rTMS)
Device: Standard rTMS (first cycle) — Patients of the SLT + STIM (standard rTMS + targeted rTMS) will firstly undergo the standard rTMS in the first 6 week of training after the baseline visit
  Arms: SLT + Brain STIM (Standard rTMS + targeted rTMS)
Device: Standard rTMS (second cycle) — Patients of the SLT + STIM (targeted rTMS + standard rTMS) will secondly undergo the standard rTMS after 12 week washout period
  Arms: Experimental: SLT + Brain STIM (targeted rTMS + Standard rTMS)
Device: Targeted rTMS (first cycle) — Patients of the SLT + STIM (targeted rTMS + standardTMS) will firstly undergo the targeted rTMS in the first 6 weeks of training after the baseline visit
  Arms: Experimental: SLT + Brain STIM (targeted rTMS + Standard rTMS)
Device: Targeted rTMS (second cycle) — Patients of the SLT + STIM (standard rTMS + targeted rTMS) will secondly undergo the targeted rTMS after 12 week washout period
  Arms: SLT + Brain STIM (Standard rTMS + targeted rTMS)

SUMMARY:
This is a monocenter randomized controlled clinical trial with cross-over arm - assessor blinded. The aims is investigating the effects of the speech language therapy (SLT) alone vs SLT + non-invasive brain stimulation (STIM), using canonic repetitive Transcranial Magnetic Stimulation (rTMS), on speech and language, clinical, neuropsychological, neuroimaging, neurophysiology, and blood features in patients with PPA.

The trial will include 45 participants suffering from semantic (svPPA), logopenic (lvPPA) or nonfluent (nfvPPA) variants of Primary Progressive Aphasia (PPA) and 30 healthy controls.

At baseline (T0) patients will undergo in-depth clinical, neuropsychological and language assessment, structural and functional magnetic resonance imaging (MRI) scan, electroencephalography (EEG) recording, functional Near Infrared Spectroscopy (fNiRS) scans, and blood sample.

PPA patients will be randomized into 2 training groups: the speech language therapy (SLT) group and the SLT + STIM (standard rTMS group or targeted rTMS).

The SLT will consist of an online intervention performed through a web-based platform. The training will be tailored to each PPA variant. svPPA and lvPPA will undergo the lexical retrieval cascade (LRC) treatment, while nfvPPA will undergo the Video-implemented Script Training (VISTA).

The SLT+ STIM group will perform the same SLT combined with non-invasive stimulation with a cross-over design: canonic repetitive Transcranial Magnetic Stimulation (rTMS) on the left dorsolateral prefrontal cortex (DLPFC) or targeted rTMS in which the site and the protocol of stimulation will be defined based on single-subject EEG combined with functional MRI (EEG+fMRI).

This design will aid in determining not only whether non-invasive stimulation can enhance clinical outcomes, but also which non-invasive stimulation is the best to improve results.

The SLT training of the SLT group will consist of 2 cycles of training lasting 1 (rest) + 5 (training) weeks, 3 times per week, 1 hour each session, separated by a 12-week washout period.

The SLT + standard or targeted STIM groups will undergo 2 cycles of 6-week training, separated by a 12-week washout period with a cross-over design: half of subjects will first receive 6-week SLT training associated with DLPFC rTMS followed by 6-week SLT associated with targeted rTMS, while the other half will follow the reverse order, according to a randomization procedure.

After the training (i.e., 6-week visit [W6] and 24-week visit [W24]), PPA patients will be re-evaluated through neurological, language, neuroimaging/neurophysiology assessments, and blood sample.

Evaluations will be also repeated at the 18-week (W18) after the wash-out and before the second cycle of treatment, as well as at 36-week (W36) and 48-week (W48) follow-up visits to assess maintenance of results. MRI and blood sample will be repeated at all visits but W18 and W36. The comprehensive neuropsychological assessment will be repeated at W48 only.

30 healthy controls will also be recruited among the spouses of patients, by word of mouth or through flyers and project awareness campaigns. They will undergo the same assessments administered to PPA patients at T0 (neurological, neuropsychological/language assessments, neuroimaging/neurophysiology, and blood sample).

Hypothesis:

1. Patients with PPA who receive a combination of SLT and rTMS will exhibit greater clinical improvement compared to those receiving SLT alone.
2. Choosing the rTMS approach and stimulation site based on individualized MRI and EEG characterization will be more effective as compared to using the standard rTMS approaches described by the literature.
3. The integration of specific clinical, cognitive, language, neuroimaging, neurophysiological, and blood features will enable the prediction of individual responses to SLT and rTMS, facilitating the development of optimized, personalized treatment plans for PPA.

DETAILED DESCRIPTION:
In the landscape of neurodegenerative disorders, neuromodulation emerges as a promising avenue for therapeutic intervention, particularly for focal neurodegenerative diseases like primary progressive aphasia (PPA). There are currently no disease-modifying drugs for PPA. Speech language training (SLT) protocols have shown some efficacy in PPA. However, the results are heterogeneous, often not sustained over time, and likely influenced by individual differences, including variations in brain reorganization. Non-invasive neuromodulation techniques, ranging from TMS to transcranial direct current stimulation, offer unique opportunities to directly influence neural activity and potentially alleviate cognitive deficits. The efficacy of such interventions, though, greatly hinges on the precision and individualization of treatment protocols. Targeted and tailored neuromodulation protocols, informed by patients' neurophysiological and structural data, could be crucial for optimizing therapeutic outcomes. By leveraging patient-specific information, such as neuroimaging and electrophysiological data, these protocols can precisely engage crucial dysfunctional neural circuits and adapt stimulation parameters to suit individual variations. In the context of PPA, where the neural substrates and symptomatology can vary widely among patients, such personalized approaches hold great promise in enhancing treatment efficacy and improving patient outcomes. Transcranial Magnetic Stimulation (TMS) has already proven to be among the most effective forms of non-invasive brain stimulation. Repetitive TMS (rTMS) of the Dorso-Lateral PreFrontal Cortex (DLPFC) has shown to be effective in PPA. Recent studies have explored the personalization of TMS treatment according to the patients' features. Here we propose a multimodal in-depth assessment that will inform precise neuro-navigated rTMS to improve functional plasticity in the most beneficial way.

PPA patients will be randomized into 2 training arms with a 1:2 ratio: the SLT group and the SLT + STIM (standard rTMS group or targeted rTMS).

Training in the SLT training will consist of 2 cycles of training lasting 1 (rest) + 5 (training) weeks, 3 times per week, 1 hour each session, separated by a 12-week washout period.

The SLT + standard or targeted STIM groups will undergo 2 cycles of 6-week training, separated by a 12-week washout period with a cross-over design: half of subjects will first receive 6-week SLT training associated with DLPFC rTMS followed by 6-week SLT associated with targeted rTMS, while the other half will follow the reverse order, according to a randomization procedure. Specifically, an induction with 20-minutes rTMS protocol for 5 consecutive days will be performed, followed by a maintenance phase where 20-minutes rTMS will be performed before each SLT session per 5 weeks, for a total of 20 rTMS sessions of whom 15 combined with SLT.

According to this design, patients will receive:

* ARM 1: 2 cycles of SLT interleaved by 12-week washout period
* ARM 2 (cross-over): 1 cycle of SLT + DLPFC rTMS and 1 cycle of SLT + targeted rTMS interleaved by 12-week washout period or viceversa.

Speech and Language Training (SLT) In all arms, the SLT intervention will be entirely administered online through a web-based platform. While each of the treatments will engage semantics, phonology, and orthography, the protocols will be tailored relative to the characteristics of each PPA variant. Patients with svPPA and lvPPA will undergo a lexical retrieval training (LRT) intervention implemented using a training cascade (Henry, et al., 2013). Patients are guided to elaborate semantic feature analysis by eliciting self-cueing retrieval strategy through identification and elaboration of spared autobiographical, semantic, orthographic, and phonological information. Participants will use noun templates to prompt themselves (e.g., What category does it belong to? What letter does the word start with? etc.). Each patient will be asked to identify and take digital photographs of items that are difficult to name but functionally relevant (e.g., related to their home life, work, hobbies). Items that will be unnamed on both two pre-treatment probes will be eligible for treatment. Stock photos of common objects will be used to supplement participant-provided items if needed. For patients with svPPA, only items with residual semantic knowledge available to the participant will be selected for treatment. The number of treatment sets will be the following: 5 items/set; 7 matched sets; two untrained sets. The target items will be trained to obtain 80% accuracy. In addition, participants will be required to complete 30 minutes of homework, at least 2 days per week, which will involve tasks similar to those completed in intervention sessions.

Patients with nfvPPA will undergo Video-implemented Script Training (VISTA), a choral reading approach training accurate production of functional scripts. The method is based on that implemented in American-English individuals with PPA and aims at improving grammar and motor aspects of speech production by taking advantage of repetitive practice and automaticity. Seven (two untrained) personalized scripts of approximately 100 words (4 sentences) each will be developed via a collaborative process between the therapist and the participant. Each script will be videotaped and will show a healthy speaker (mouth only) producing each script. Articulatory gestures will be exaggerated to provide salient visual cues for production. Syntactic and articulatory difficulty of scripts and rate of speech for videos will be tailored to each participant. Participants will receive immediate feedback regarding production, with an emphasis on grammatical correctness as well as articulator placement and speech sound accuracy. The target scripts will be trained until they are produced with 90% accuracy over two sessions. Patients will be asked to complete 30 minutes of daily homework (oral reading practice with sentences presented visually and auditorily via a recordable photo album). Treatment probes will be taken at the beginning of each session, comprising a request for information on each script topic (trained and untrained). The overall final schedule for all patients will be one set/script reviewed per session, 3 one-hour sessions/week for 5 weeks.

Non-Invasive Brain Stimulation (rTMS) For the SLT + standard STIM group, we will treat patients by stimulating the Left DorsoLateral Prefrontal Cortex (DLPFC); rTMS will be administered as high-frequency (20Hz) in 2 second trains (40 pulses per train) with an inter-train interval of 22 seconds for a total of 50 trains (2000 pulses per session) at 120% of the patient's resting motor threshold. Patients will undergo an induction with 20-minutes rTMS protocol for 5 consecutive days, then they will start a maintenance phase where rTMS will be performed 3 days a week per 20 minutes preceding the SLT session, for a total of 20 sessions (of whom 15 combined with SLT).

For the SLT + targeted STIM group, the protocol will be the same, but the site of stimulation will be defined using EEG/fMRI recordings of language tasks (syntax production for nfvPPA; silent naming for svPPA and lvPPA) to evidence the areas of higher activation/connectivity of the language network. We will define the area of higher fMRI activation; then, we will use fMRI-EEG connectivity and spectral activity to select the site of stimulation, among the areas with the highest fMRI activation and the highest Beta/Gamma frequencies.

Additional procedure will be language evaluation, neuroimaging/neurophysiology (EEG, MRI, fNiRS, EEG/fMRI of language tasks) acquisitions, and blood sample.

Follow-up assessments will be performed at the San Raffaele Neurotech Hub, UniSR.

At each follow-up timepoint (W6, W18, W24, W36 and W48) patients will repeat the following evaluations:

1. Neurological evaluation: Clinical Dementia Rating-Frontotemporal dementia (CDR-FTD) for assessing disease severity, basic and instrumental activities of daily life (ADL and IADL) for assessing independency, mini mental state examination (MMSE) and frontal assessment battery (FAB) for assessing global cognition.
2. Speech and Language assessment: a quantitative assessment of the correct naming of trained and untrained items for patients undergoing the LRC treatment (lvPPA/svPPA), changes in percentage of VISTA script words produced correctly for trained and untrained scripts (nfvPPA), and changes in Patient and Caregiver Self-Rating using ad hoc scale of Communication Effectiveness and the Italian version of the Communication Outcome after Stroke scale (COAST) (all PPA) will be performed. To analyze the connected speech, we will use the Nicholas and Brookshire (1993) picture description task and the report of a relevant event; with using these samples, we will calculate correct information unit (IU), in order to examine informativeness and efficiency of communication. Speech samples will also be analyzed for number of grammatically completed utterances (presence of appropriate agent, verb, and patient). A comprehensive language testing will further include the examination of: verb and sentence production with the Italian version of the Northwestern Assessment of Verbs and Sentences (NAVS-I); confrontation naming and single-word comprehension with the naming and word picture matching subtests, respectively, of the CaGi battery; object knowledge with the Semantic Association Task; comprehension of syntactically complex sentences with the syntax comprehension test; syntax production with the Italian version of the Northwestern Anagram Test (NAT-I); word and sentence repetition with the subtest of the Aachener Aphasie Test (AAT), and word and non-word repetition with the subtest of the ENPA; fluency with the phonemic and semantic fluency tests; motor speech with an unpublished scale. The screening for Aphasia in Neurodegeneration (SAND) will be also administered.
3. Neurophysiology (EEG): All participants will undergo prolonged 64-channels EEG recording. EEGs will be recorded in a quiet room with dimmed lights. Electrodes are placed according to the extended 10-20 system using a pre-cabled head set. Electrode impedance is below 5 KΩ. As reference, bilateral mastoid bone electrodes will be used. The ground electrode will be Fz. The sampling rate will be set at 256 Hz; A/D conversion is made at 16 bits; the pre-amplifiers amplitude range is ±3200 μV. Hardware acquisition filters are used: high pass = 0.2 Hz; low-pass = 128 Hz. We will record 2 separate conditions: resting Eyes Closed and Resting Eyes open.
4. Neuroimaging (fNiRS): fNiRS will be used to record the continuous spectral wave of brain resting activity. The acquisition time will last 10 minutes, to include at least five low frequency periods (0.01 Hz) to ensure the effectiveness of subsequent phase-related analysis. The subjects will be asked to sit quietly on a stool with armrests facing the same direction in the same room, staying relaxed and ensuring that they are awake to avoid falling asleep. The optometer head-set will comprise 8 light sources and 8 probes, which will be arranged in the left and right hemisphere following the 10-20 montage. The sampling frequency is set to 10 Hz using two wavelengths (760 nm and 850 nm) for scanning.

At W6, W24 and W48 patients will perform also:

Neuroimaging (brain MRI): T2-weighted spin echo to exclude cerebrovascular alterations; three-dimensional (3D) sagittal T1-weighted fast field echo to assess grey matter alterations; T2*-weighted EP imaging (EPI) sequence for resting state fMRI; axial pulsed-gradient spin echo (PGSE) single shot DW EPI sequence for white matter alterations.

Blood sample: A blood draw will be performed (20 ml). From the collected blood sample, plasma will be separated, which will be used for the specific analysis of serum NfL.

At W48 patients will perform also:

Neuropsychological assessment: standard and comprehensive cognitive evaluation assessing all the cognitive domains (memory, executive functions, attention, visuo-spatial abilities, social cognition, language), mood and behaviour.

According to study design, the end of the study is defined as the date of completion of any study-related analysis.

ELIGIBILITY:
Inclusion Criteria for patients

* Clinical and imaging-supported diagnosis of any variant of PPA (svPPA, lvPPA, nfvPPA) according to international diagnostic criteria (Gorno- Tempini et al., 2011)
* Age range: 40-85
* MMSE>15
* Native Italian Speaker
* Right handedness
* Stable pharmacological treatment of at least 4 weeks and without any change during the observation period (48 weeks)
* Oral and written informed consent to study participation

Exclusion Criteria for patients

* Any major systemic, psychiatric, neurological, and visual disturbance
* Medical conditions or substance abuse that could interfere with cognition
* Hypoacusis or severe visual deficits
* Pacemaker and/or other implanted neurostimulation devices in the head/neck district
* (Other) Contraindications to undergoing MRI examination
* Brain damage at routine MRI, including extensive cerebrovascular disorders
* Denied oral and written informed consent to study participation
* Inability to repeat multisyllabic words (4 syllables)
* Concomitant participation to other pharmacological and non pharmacological studies
* Traumatic or surgical wounds that could determine a risk of infection in the site of non-invasive stimulation
* Scalp alterations that could determine the spread of excessive current from the device.
* Known history of epilepsy (due to small risk of seizure induction from rTMS in epileptic patients

Inclusion criteria for healthy controls:

* Sex-matched and age-matched (age range: mean age of PPA years ± 15 years)
* MMSE>27
* Native Italian Speaker
* Right handedness
* Oral and written informed consent to study participation

Exclusion criteria for healthy controls:

* Any major systemic, psychiatric, neurological, and visual disturbance
* Medical conditions or substance abuse that could interfere with cognition
* Hypoacusis or severe visual deficits
* Pacemaker and/or other implanted neurostimulation devices in the head/neck district
* (Other) Contraindications to undergoing MRI examination
* Brain damage at routine MRI, including extensive cerebrovascular disorders
* Denied oral and written informed consent to study participation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Changes in number of correct naming of trained items for patients lvPPA undergoing LRC alone vs LRC + STIM treatment | Baseline, week 6, week 24
  The primary objective is assessing the effect of SLT alone vs SLT + STIM (standard and targeted rTMS) on PPA speech and language features.
  This will be measured trough the primary endpoint regarding changes in number of correct naming of trained items for lvPPA patients undergoing the LRC alone vs LRC + STIM treatment
Changes in number of correct naming of trained items for patients svPPA undergoing LRC alone vs LRC+STIM treatment | Baseline, week 6, week 24
  The primary objective is assessing the effect of SLT alone vs SLT + STIM (standard and targeted rTMS) on PPA speech and language features.
  This will be measured trough the primary endpoint regarding changes in number of correct naming of trained items for svPPA patients undergoing the LRC alone vs LRC + STIM treatment
Changes in Percentage of VISTA script words produced correctly for trained scripts for nfvPPA patients undergoing VISTA alone vs VISTA + STIM treatment | Baseline, week 6, week 24
  The primary objective is assessing the effect of SLT alone vs SLT + STIM (standard and targeted rTMS) on PPA speech and language features.
  This will be measured trough the primary endpoint regarding changes in percentage of VISTA words produced correctly for trained scripts for nfvPPA patients undergoing VISTA alone vs VISTA + STIM treatment
Measures of Patient and Caregiver Self-Rating of Communication Effectiveness in all PPA patients undergoing LST alone vs LST + STIM | Baseline, week 6, week 24
  The primary objective is assessing the effect of SLT alone vs SLT + STIM (standard and targeted rTMS) on PPA speech and language features. This will be measured trough the primary endpoint regarding Measures of Patient and Caregiver Self-Rating of Communication Effectiveness in all PPA patients undergoing SLT alone vs SLT + STIM treatment

SECONDARY OUTCOMES:
Changes in number of correct naming of trained items for patients lvPPA undergoing the LRC + STIM treatment , according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is assessing the effects of two different modalities of non-invasive stimulation (standard vs targeted rTMS) along with SLT treatment on lvPPA patients' speech and language features. This will be evaluated trough the secondary endpoint regarding changes in number of correct naming of trained items for patients lvPPA undergoing the LRC + STIM treatment , according to the cross-over design (LRC + standard rTMS vs LRC + targeted rTMS)
Changes in number of correct naming of trained items for patients svPPA undergoing the LRC + STIM treatment , according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is assessing the effects of two different modalities of non-invasive stimulation (standard vs targeted rTMS) along with SLT treatment on svPPA patients' speech and language features. This will be evaluated trough the secondary endpoint regarding changes in number of correct naming of trained items for patients svPPA undergoing the LRC + STIM treatment , according to the cross-over design (LRC + standard rTMS vs LRC + targeted rTMS)
Changes in Percentage of VISTA script words produced correctly for trained scripts for nfvPPA patients undergoing the VISTA + STIM treatment, according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is assessing the effects of two different modalities of non-invasive stimulation (standard vs targeted rTMS) along with SLT treatment on nfvPPA patients' speech and language features. This will be evaluated trough the secondary endpoint regarding changes in percentage of VISTA script words produced correctly for trained scripts for nfvPPA patients undergoing the VISTA + STIM treatment, according to the cross-over design (VISTA + standard rTMS vs VISTA+ targeted rTMS)
Measures of Patient and Caregiver Self-Rating of Communication Effectiveness (all PPA) undergoing SLT + STIM treatment, according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is assessing the effects of two different modalities of non-invasive stimulation (standard vs targeted rTMS) along with LST treatment on all PPA patients' speech and language features. This will be evaluated trough the secondary endpoint regarding Measures of all PPA Patient and Caregiver Self-Rating of Communication Effectiveness in all PPA patients undergoing LST + STIM treatment, according to the crossover design (LST + standard rTMS vs LST + targeted rTMS).
Changes in number of correct naming of untrained items for lvPPA patients undergoing LRC alone vs LRC + STIM treatment | Baseline, week 6, week 24
  The secondary objective is also evaluating the generalization of clinical benefits of SLT alone vs SLT+ STIM treatment.This objective can be evaluated trough the secondary endpoint regarding the patient's improvement in retrieving words that were not directly trained with the therapist during LRC treatment. If the patient improves in the retrieval of words not directly trained, it means that the treatment has enhanced the mechanisms of vocabulary access. going beyond simple repetition of the words practiced. Thus, the outcome for this objective is changes in number of correct naming of untrained items for patients lvPPA undergoing the LRC alone vs LRC + STIM treatment
Changes in number of correct naming of untrained items for svPPA patients undergoing LRC alone vs LRC + STIM treatment | Baseline, week 6, week 24
  The secondary objective is also evaluating the generalization of clinical benefits of SLT alone vs SLT+ STIM treatment.This objective can be evaluated trough the secondary endpoint regarding the patient's improvement in retrieving words that were not directly trained with the therapist during LRC treatment. If the patient improves in the retrieval of words not directly trained, it means that the treatment has enhanced the mechanisms of vocabulary access. going beyond simple repetition of the words practiced. Thus, the outcome for this objective is changes in number of correct naming of untrained items for patients svPPA undergoing the LRC alone vs LRC + STIM treatment
Changes in percentage of VISTA script words produced correctly for untrained scripts for nfvPPA patients undergoing VISTA alone vs VISTA + STIM treatment | Baseline, week 6, week 24
  The secondary objective is also evaluating the generalization of clinical benefits of SLT alone vs SLT+ STIM treatment. This objective can be evaluated trough the secondary endpoint regarding the patient's improvement in producing correctly words for new scripts that were not directly trained with the therapist during VISTA treatment. This means that the patient is not only improving in the specific trained scripts but also in broader speech production. Thus, the primary outcome for this objective is changes in percentage of VISTA script words produced correctly for untrained scripts for nfvPPA patients undergoing VISTA alone vs VISTA + STIM treatment
Changes in number of correct naming of untrained items for patients lvPPA undergoing the LRC + STIM treatment according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is also evaluating the generalization of clinical benefits of SLT+ STIM treatment, according to the crossover design (SLT + standard rTMS vs SLT + targeted rTMS). This objective can be evaluated trough the secondary endpoint regarding the patient's improvement in retrieving words that were not directly trained with the therapist during LRC treatment. If the patient improves in the retrieval of words not directly trained, it means that the treatment has enhanced the mechanisms of vocabulary access. going beyond simple repetition of the words practiced. Thus, the outcome for this objective is changes in number of correct naming of untrained items for patients lvPPA undergoing the LRC + STIM treatment according to the cross-over design (LRC + standard rTMS vs LRC + targeted rTMS)
Changes in number of correct naming of untrained items for patients svPPA undergoing the LRC + STIM treatment according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is also evaluating the generalization of clinical benefits of SLT + STIM according to the crossover design (SLT + standard rTMS vs SLT + targeted rTMS). This objective can be evaluated trough the secondary endpoint regarding the patient's improvement in retrieving words that were not directly trained with the therapist during LRC treatment. If the patient improves in the retrieval of words not directly trained, it means that the treatment has enhanced the mechanisms of vocabulary access. going beyond simple repetition of the words practiced. Thus, the outcome for this objective is changes in number of correct naming of untrained items for patients svPPA undergoing the LRC + STIM treatment according to the cross-over design (LRC + standard rTMS vs LRC + targeted rTMS)
Changes in Percentage of VISTA script words produced correctly for untrained scripts, for nfvPPA patients undergoing VISTA + STIM treatment, according to the cross-over design (standard vs targeted rTMS) | Baseline, week 6, week 24
  The secondary objective is also evaluating the generalization of clinical benefits of SLT + STIM treatment, according to the crossover design (SLT + standard rTMS vs SLT + targeted rTMS) This objective can be evaluated trough the secondary endpoint regarding the patient's improvement in producing correctly words for new scripts that were not directly trained with the therapist during VISTA treatment. This means that the patient is not only improving in the specific trained scripts but also in broader speech production. Thus, the primary outcome for this objective is changes in percentage of VISTA script words produced correctly for untrained scripts for nfvPPA patients undergoing VISTA + STIM treatment according to the cross-over design (VISTA + standard rTMS vs VISTA+ targeted rTMS)
Changes in number of correct items for lvPPA patients undergoing the LRC alone vs LRC + STIM | Week 6, Week 18, Week 24, Week 36, Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT alone vs SLT+ STIM treatment. This objective will be evaluated trough the secondary outcome regarding changes in number of correct naming of trained items for lvPPA patients undergoing LRC alone vs LRC + STIM treatment
Changes in number of correct items for svPPA patients undergoing the LRC alone vs LRC + STIM | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT alone vs SLT + STIM treatment. This objective will be evaluated trough the secondary outcome regarding changes in number of correct naming of trained items for svPPA patients undergoing LRC alone vs LRC + STIM treatment
Changes in Percentage of VISTA script words produced correctly for trained scripts for nfvPPA patients undergoing VISTA alone vs VISTA + STIM | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT alone vs SLT + STIM treatment. This objective will be evaluated trough the secondary outcome regarding changes in percentage of VISTA script words produced correctly for trained scripts in nfvPPA patients undergoing VISTA alone vs VISTA + STIM treatment
Changes in number of correct naming of trained items for lvPPA patients undergoing LRC + STIM treatment, according to the crossover design (standard rTMS vs targeted rTMS) | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT according to the crossover design (SLT + standard rTMS vs SLT + targeted rTMS). This objective will be evaluated trough the secondary outcome regarding changes in number of correct naming of trained items for lvPPA patients undergoing the LRC + STIM treatment, according to the crossover design (LRC + standard rTMS vs LRC + targeted rTMS)
Changes in number of correct naming of trained items for svPPA patients undergoing LRC + STIM treatment, according to the crossover design (standard rTMS vs targeted rTMS) | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT according to the crossover design (SLT + standard rTMS vs SLT + targeted rTMS). This objective will be evaluated trough the secondary outcome regarding changes in number of correct naming of trained items for svPPA patients undergoing the LRC + STIM treatment, according to the crossover design (LRC + standard rTMS vs LRC + targeted rTMS)
Changes in Percentage of VISTA script words produced correctly for trained scripts for nfvPPA patients undergoing VISTA + STIM treatment, according to the crossover design (standard rTMS vs targeted rTMS) | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT according to the crossover design (SLT + standard rTMS vs SLT + targeted rTMS). This objective will be evaluated trough the secondary outcome regarding changes in percentage of VISTA script words produced correctly for trained scripts in nfvPPA patients undergoing VISTA + STIM treatment, according to the crossover design (VISTA + standard rTMS vs VISTA+ targeted rTMS)
Measures of Patient and Caregiver Self-Rating of Communication Effectiveness in all PPA patients undergoing SLT alone vs SLT+ STIM treatment | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT alone vs SLT+ STIM treatment. This objective will be evaluated trough Measures of Patient and Caregiver Self-Rating of Communication Effectiveness in all PPA patients undergoing SLT alone vs SLT+ STIM treatment
Measures of Patient and Caregiver Self-Rating of Communication Effectiveness for all PPA patients undergoing SLT +STIM treatment, according to the crossover design | Week 6, Week 18, Week 24, Week 36 and Week 48
  The secondary objective is also evaluating the maintenance of clinical benefits of SLT + STIM, according to the two stimulation modalities (standard vs targeted rTMS) in all PPA. This objective will be evaluated trough Measures of Patient and Caregiver Self-Rating of Communication Effectiveness in all PPA patients undergoing SLT + STIM, according to the crossover design

OTHER OUTCOMES:
Changes in cognitive measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline, Week 6, Week18, Week24, Week36, Week48
  The objective is evaluating the effects of SLT vs SLT + STIM on cognitive features like accuracy (number of correct answer) in global cognition, memory, attention and executive functions, visuospatial abilities and social cogntion.
  This will be evaluated trough neuropsychological test battery
Changes in cognitive measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM ,according to the crossover design, on cognitive features like accuracy (number of correct answer) in global cognition, memory, attention and executive functions, visuospatial abilities and social cogntion. This will be evaluated trough neuropsychological test battery
Changes in language measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline, Week 6, Week18, Week24, Week36, Week48
  The objective is evaluating the effects of SLT vs SLT + STIM on language features like accuracy (number of correct answers) and/or latency (time for completing the task) in connected speech, syntax production and comprehension, motor speech, verbal repetition, writing and reading, naming and single-word comprehension, semantic knowledge. This will be evaluated trough Nicholas and Brookshire picture for assessing efficiency of communication; Northwestern Anagram Test (NAT-I) and Northwestern Assessment of Verbs and Sentences (NAVS-I) for Italian for assessing syntax production; Italian syntax comprehension for assessing syntax comprehension; Motor Speech Evaluation Scale for assessing motor speech; Aachener Aphasie Test (AAT) and the ENPA battery for assessing verbal repetition; AAT for assessing writing and reading; CaGi battery for assessing naming and single-word comprehension; Semantic Association Task (SAT) and the Pyramids and Palm Trees Test for assessing semantic knowledge.
Changes in language measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM according to the crossover design on language features like accuracy (number of correct answers) and/or latency (time for completing the task) in connected speech, syntax production and comprehension, motor speech, verbal repetition, writing and reading, naming and single-word comprehension, semantic knowledge. This will be evaluated trough Nicholas and Brookshire picture for assessing efficiency of communication; Northwestern Anagram Test (NAT-I) and Northwestern Assessment of Verbs and Sentences (NAVS-I) for Italian for assessing syntax production; Italian syntax comprehension for assessing syntax comprehension; Motor Speech Evaluation Scale for assessing motor speech; Aachener Aphasie Test (AAT) and the ENPA battery for assessing verbal repetition; AAT for assessing writing and reading; CaGi battery for assessing naming and single-word comprehension; Semantic Association Task (SAT) and the Pyramids and Palm Trees Test
Changes in MRI measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline, Week 6, Week 18, Week 24, Week 36, Week 48
  The objective is evaluating the effects of SLT vs SLT + STIM on MRI features like gray matter volumes and thickness; changes in BOLD signal; white matter microstructure integrity.
  This will be evaluated trough three-dimensional (3D) sagittal T1-weighted fast field echo for assessing grey matter alterations; T2*-weighted EP imaging (EPI) sequence for resting state functional MRI to assess changes in BOLD signal; axial pulsed-gradient spin echo (PGSE) single shot DW EPI sequence for assessing white matter microstructural alterations.
Changes in MRI measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) on MRI features like gray matter volumes and thickness; changes in BOLD signal; white matter microstructure integrity. This will be evaluated trough three-dimensional (3D) sagittal T1-weighted fast field echo for assessing grey matter alterations; T2*-weighted EP imaging (EPI) sequence for resting state functional MRI to assess changes in BOLD signal; axial pulsed-gradient spin echo (PGSE) single shot DW EPI sequence for assessing white matter microstructural alterations.
Changes in EEG measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline , Week 6, Week 18, Week 24, Week 36, Week 48
  The objective is evaluating the effects of SLT vs SLT + STIM on EEG features in PPA patients. EEG will be analyzed in the frequency domain using Power Spectral Analysis, in the connectivity domain using WPLI and various methods for the quantification of topological graph theory metrics. Finally, other metrics such as entropy and signal complexity will be used
Changes in EEG measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) on EEG features in PPA patients. EEG will be analyzed in the frequency domain using Power Spectral Analysis, in the connectivity domain using WPLI and various methods for the quantification of topological graph theory metrics. Finally, other metrics such as entropy and signal complexity will be used
Changes in FNiRS measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline, week 6, week 18, week 24, week 36, week 48
  The objective is evaluating the effects of SLT vs SLT + STIM on fNiRS features like concentration of hemoglobin (blood oxygenation) changes. This will be evaluated trough near-infrared light spectroscopy
Changes in FNiRS measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) on fNiRS features like concentration of hemoglobin (blood oxygenation) changes. This will be evaluated trough near-infrared light spectroscopy
Changes in blood measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline, week 6, week 18, week 24, week 36, week 48
  The objective is evaluating the effects of SLT vs SLT + STIM on blood features like Serum neurofilaments (NfL), Aβ42, Aβ40, pTau-181 and pTau-217 levels. A blood draw will be performed (20 ml).
Changes in blood measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) on blood features like Serum neurofilaments (NfL), Aβ42, Aβ40, pTau-181 and pTau-217 levels. A blood draw will be performed (20 ml).
Changes in clinical measures in PPA patients undergoing SLT alone vs SLT + STIM treatment | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT vs SLT + STIM on clinical features like disease diversity and indipendence. This will be evaluated trough Clinical Dementia Rating-Frontotemporal dementia (CDR-FTD) for assessing disease severity, basic and instrumental activities of daily life (ADL and IADL) for assessing independence.
Changes in clinical measures in PPA patients undergoing SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) | Baseline, Week 6, Week 18, Week 24, Week 36 and Week 48
  The objective is evaluating the effects of SLT + STIM according to the crossover design (standard rTMS vs targeted rTMS) on clinical features like disease diversity and indipendence. This will be evaluated trough Clinical Dementia Rating-Frontotemporal dementia (CDR-FTD) for assessing disease severity, basic and instrumental activities of daily life (ADL and IADL) for assessing independence.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Massimo Filippi, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- San Raffaele Neurotech Hub, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No